CLINICAL TRIAL: NCT00238329
Title: Phase II Study of Pegylated Interferon and Thalidomide in Pretreated Metastatic Malignant Melanoma
Brief Title: PEG-Interferon Alfa-2b and Thalidomide in Treating Patients With Recurrent or Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445593; P30CA022453 (NIH); WSU-C-2257; WSU-HIC-120900M01-FB
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; iris melanoma; recurrent intraocular melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — peginterferon alfa-2b; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: PEG-interferon alfa-2b
Drug: thalidomide

SUMMARY:
RATIONALE: PEG-interferon alfa-2b may interfere with the growth of tumor cells. Biological therapies, such as thalidomide, may stimulate the immune system in different ways and stop tumor cells from growing. PEG-interferon alfa-2b and thalidomide may also stop the growth of melanoma by blocking blood flow to the tumor. Giving PEG-interferon alfa-2b together with thalidomide may be an effective treatment for melanoma.

PURPOSE: This phase II trial is studying how well giving PEG-interferon alfa-2b together with thalidomide works in treating patients with recurrent or metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with recurrent or metastatic malignant melanoma treated with PEG-interferon alfa-2b and thalidomide.
* Determine the quantitative and qualitative toxic effects of this regimen in these patients.
* Determine progression-free and overall survival of patients treated with this regimen.

OUTLINE: Patients receive PEG-interferon alfa-2b subcutaneously once weekly and oral thalidomide once daily. Treatment continues for at least 2 weeks but no more than 8 months in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive PEG-interferon alfa-2b and thalidomide for 2 months beyond documentation of CR.

PROJECTED ACCRUAL: A total of 18-32 patients will be accrued for this study within 14-38 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma, including any of the following:

  * Cutaneous melanoma
  * Ocular melanoma
  * Mucosal melanoma
  * Unidentified primary tumor
* Recurrent or metastatic disease
* Bidimensionally measurable or evaluable disease
* Brain metastases allowed provided disease is stable for ≥ 6 weeks after prior radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* SWOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* SGOT ≤ 2 times ULN

Renal

* Creatinine ≤ 2 mg/dL

Cardiovascular

* None of the following conditions within the past 3 months:

  * Congestive heart failure
  * Second- or third-degree heart block
  * Myocardial infarction

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception (1 highly effective and 1 additional method) for ≥ 4 weeks before, during, and for ≥ 4 weeks after completion of study treatment
* No other malignancy within the past 2 years except adequately treated skin cancer or carcinoma in situ of the cervix
* No concurrent blood, sperm, or ova donation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior biologic therapy (e.g., interferon) allowed

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 28 days since prior radiotherapy

Surgery

* At least 28 days since prior surgery

Other

* No more than 2 prior systemic treatment regimens for metastatic malignant melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2001-01; Primary Completion 2005-12 (Actual); Study Completion 2007-06

PRIMARY OUTCOMES:
Response rate as measured scans and tumor measurements every 8 weeks
Qualitative and quantitative toxicities at 30 days following study treatment

SECONDARY OUTCOMES:
Progression-free survival by standard life table and Kaplan-Meier
Overall survival by standard life table and Kaplan-Meier
Vascular flow to metastatic sites by positron-emission tomography scan every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulka N. Vaishampayan, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States